CLINICAL TRIAL: NCT01486550
Title: Effect of Hydroxyethyl Starch on Renal Handling of Salt and Water, Blood Pressure-regulating Hormones, Proteins and Circulatory System of Patients Undergoing Kidney Removal by Keyhole Surgery
Brief Title: Hydroxyethyl Starch and Renal Function After Laparoscopic Nephrectomy
Acronym: VONE
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of patient enrollment
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ASK-1-2011
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — HES 130-0.4; Hydroxyethyl Starch Derivatives; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voluven (Hydroxyethyl starch 130/0,4) (Active Comparator): Patients undergoing laparoscopic nephrectomy will receive either fluid therapy with active comparator (Voluven) or placebo (Sodium Chloride)
  Interventions: Drug: Voluven (Hydroxyethyl starch 130/0,4)
- Sodium Chloride 9mg/ml (Placebo Comparator): Patients undergoing laparoscopic nephrectomy will receive either fluid therapy with active comparator (Voluven) or placebo (Sodium Chloride)
  Interventions: Drug: Sodium Chloride 9mg/ml

INTERVENTIONS:
Drug: Voluven (Hydroxyethyl starch 130/0,4) — 7,5 ml/kg in the first hour and then 5 ml/kg minimum
  Other Names: Voluven; Hydroxyethyl starch; Venofundin
  Arms: Voluven (Hydroxyethyl starch 130/0,4)
Drug: Sodium Chloride 9mg/ml — 7,5 ml/kg in the first hour and then 5 ml/kg
  Other Names: Isotone saline solution
  Arms: Sodium Chloride 9mg/ml

SUMMARY:
The purpose of this project is to investigate if hydroxyethyl starch (HES) is potential nephrotoxic and examine the effects on the circulation and kidneys during administration of HES during surgery.

DETAILED DESCRIPTION:
Hydroxyethyl starch (HES) is widely used in hospitals to maintain circulation in critically ill patients. In recent years studies have raised suspicion that HES is nephrotoxic. So far acute kidney injury has been diagnosed based on creatinine measurements, but new technology allows for earlier diagnosis using measurements of biomarkers in urine. The purpose of this project is to investigate HES's potential toxicity and effects on the circulation and kidneys using measurements of biomarkers specific for toxicity and for the sodium/water balance in the urine and by measurements of vasoactive hormones in the blood after administration of HES 130/0.4

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Males and females
* Indication for laparoscopic nephrectomy

Exclusion Criteria:

* Blood donation within the last month
* Lack of wish to participate
* eGFR< 15ml/min
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-12; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
u-NGAL | 2-4 hours
  The main objective for the trial(only patients undergoing elective laparoscopic nephrectomy) is to measure the effect of hydroxyethyl starch on u-NGAL, which is a biomarker of nephrotoxicity

SECONDARY OUTCOMES:
u-Kim1 and u-LFABP | 2-4 hours
  Another objective for the trial(only patients undergoing elective laparoscopic nephrectomy) is to measure the effect of hydroxyethyl starch on u-Kim1 and u-LFAPB, which are also biomarkers of nephrotoxicity
FENa, u-ENaCβ, CH2O, u-AQP2,u-NCC, u-NK2CC | 2-4 hours
  Secondarily to measure the effect of hydroxyethyl starch on the renal tubular transport of sodium and water during elective laparoscopic nephrectomy
PRC, p-Ang-II, p -Aldo, p-ANP,P-GDP, p-AVP, p-Endothelin | 2-4 hours
  Thirdly to measure the effect of hydroxyethyl starch on vasoactive hormones during elective laparoscopic nephrectomy
SBP, DBP, heartrate | 2-4 hours
  Fourthly measure the effect of hydroxyethyl starch on central hemodynamics during elective laparoscopic nephrectomy

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sophie P. Kancir, MD PhD, Principal Investigator — Regional Hospital Holstebro
Locations (1):
- Medicinck forskningsafsnit, Regionshospitalet Holstebro, Holstebro, Denmark